CLINICAL TRIAL: NCT00869661
Title: A Randomized, Double-blind, Multicenter, Dose and Duration Finding Study to Evaluate the Sustained Virologic Response of the HCV Polymerase Inhibitor Prodrug (RO5024048) in Combination With Pegasys® and Ribavirin® (SOC) Versus SOC in Treatment-Naïve Patients With HCV Genotype 1 or 4 Infection
Brief Title: A Study of RO5024048 in Combination With Pegasys and Copegus in Treatment-Naive Patients With Chronic Hepatitis C, Genotype 1 or 4
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NV20536; 2008-008258-21
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin; peginterferon alfa-2a

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- Group 1 (Experimental): RO5024048 500 mg bid + Pegasys + Copegus for 12 weeks, followed by SOC for 12 weeks. After 24 weeks, patients who have achieved rapid viral response will stop treatment, and those who have not will receive SOC for a further 24 weeks.
  Interventions: Drug: Copegus; Drug: Pegasys; Drug: RO5024048
- Group 2 (Experimental): RO5024048 1000mg bid + Pegasys + Copegus for 8 weeks, followed by SOC for 16 weeks. After 24 weeks, patients who have achieved rapid viral response will stop treatment, and those who have not will receive SOC for a further 24 weeks.
  Interventions: Drug: Copegus; Drug: Pegasys; Drug: RO5024048
- Group 3 (Experimental): RO5024048 1000mg bid + Pegasys + Copegus for 12 weeks, followed by SOC for 12 weeks. After 24 weeks, patients who have achieved rapid viral response will stop treatment, and those who have not will receive SOC for a further 24 weeks.
  Interventions: Drug: Copegus; Drug: Pegasys; Drug: RO5024048
- Group 4 (Experimental): Group 4 will receive RO5024048 1000mg bid + Pegasys + Copegus for 12 weeks, followed by SOC for 36 weeks
  Interventions: Drug: Copegus; Drug: Pegasys; Drug: RO5024048
- Group 5 (Active Comparator): Group 5 will receive SOC for 48 weeks
  Interventions: Drug: Copegus; Drug: Pegasys
- Group 6 (Experimental): Group 6 provides retreatment on an open-label basis for patients of Group 5 who failed treatment. Patients will receive RO5024048 1000mg bid + Pegasys + Copegus for 24 weeks, followed by SOC for 24 weeks.
  Interventions: Drug: Copegus; Drug: Pegasys; Drug: RO5024048

INTERVENTIONS:
Drug: Copegus — 1000/1200mg po daily for 24 or 48 weeks
  Arms: Group 1; Group 2; Group 3
Drug: Copegus — 1000/1200mg po daily for 48 weeks
  Arms: Group 4; Group 5; Group 6
Drug: Pegasys — 180 micrograms sc weekly for 24 or 48 weeks
  Arms: Group 1; Group 2; Group 3
Drug: Pegasys — 180 micrograms sc weekly for 48 weeks
  Arms: Group 4; Group 5; Group 6
Drug: RO5024048 — 1000mg bid for 24 weeks
  Arms: Group 6
Drug: RO5024048 — 500mg bid for 12 weeks
  Arms: Group 1
Drug: RO5024048 — 1000mg bid for 8 weeks
  Arms: Group 2
Drug: RO5024048 — 1000mg bid for 12 weeks
  Arms: Group 3; Group 4

SUMMARY:
This 6-arm study will assess the efficacy and safety of RO5024048 (R7128) in combination with the approved doses of Pegasys (180micrograms sc weekly) + Copegus (1000/1200mg po daily) (SOC), versus SOC in treatment-naive patients with chronic hepatitis C, genotype 1 and 4. The first 3 groups will receive 1) RO5024048 500mg bid + Pegasys + Copegus for 12 weeks, followed by SOC for 12 weeks; 2)RO5024048 1000mg bid + Pegasys + Copegus for 8 weeks, followed by SOC for 16 weeks; 3) RO5024048 1000mg bid + Pegasys + Copegus for 12 weeks, followed by SOC for 12 weeks. After 24 weeks, patients in these 3 groups who have achieved rapid viral response will stop treatment, and those who have not will receive SOC for a further 24 weeks. Group 4 will receive RO5024048 1000mg bid + Pegasys + Copegus for 12 weeks, followed by SOC for 36 weeks, and group 5 will receive SOC for 48 weeks. Group 6 provides retreatment on an open-label basis for patients of Group 5 who failed treatment. Patients will receive RO5024048 1000mg bid + Pegasys + Copegus for 24 weeks, followed by SOC for 24 weeks. The anticipated time on study treatment is 6-12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 18-65 years of age
* Chronic hepatitis C, genotype 1 or 4
* Treatment-naive

Exclusion Criteria:

* No previous treatment with any interferon- or ribavirin-based therapy
* Other forms of liver disease
* HIV infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2001-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Sustained virologic response: Percentage of patients with undetectable Hepatitis C RNA level | 24 weeks after end of treatment

SECONDARY OUTCOMES:
Virologic response: Percentage of patients with undetectable Hepatitis C RNA level | 60 Weeks
Virologic response: Percentage of patients with undetectable Hepatitis C RNA level | 12 weeks post-treatment
Relapse rate: Percentage of patients who achieved a virologic response at the end of treatment but had detectable Hepatitis C RNA level at the last assessment post treatment | 72 weeks
Safety: Incidence of adverse events | 72 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (62):
- United States (21):
  - Birmingham, Alabama
  - La Jolla, California
  - Sacramento, California
  - San Diego, California
  - San Francisco, California
  - Washington D.C., District of Columbia
  - Bradenton, Florida
  - Gainesville, Florida
  - Marietta, Georgia
  - Chicago, Illinois
  - Lutherville, Maryland
  - Kansas City, Missouri
  - Newark, New Jersey
  - New York, New York
  - Hershey, Pennsylvania
  - Providence, Rhode Island
  - Columbia, South Carolina
  - Nashville, Tennessee
  - Houston, Texas
  - San Antonio, Texas
  - Richmond, Virginia
- Australia (8):
  - Sydney, New South Wales
  - Greenslopes, Queensland
  - Herston, Queensland
  - Woolloongabba, Queensland
  - Fitzroy, Victoria
  - Melbourne, Victoria
  - Nedlands, Western Australia
  - Perth, Western Australia
- Vienna, Austria
- Canada (6):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - London, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- France (7):
  - Créteil
  - La Tronche
  - Lille
  - Nice
  - Paris
  - Pessac
  - Vandœuvre-lès-Nancy
- Germany (6):
  - Berlin
  - Frankfurt am Main
  - Freiburg im Breisgau
  - Hanover
  - München
  - Ulm
- Italy (4):
  - Bologna, Emilia-Romagna
  - Milan, Lombardy
  - Turin, Piedmont
  - Pisa, Tuscany
- Santurce, Puerto Rico
- Spain (7):
  - Badalona, Barcelona
  - Barcelona, Barcelona
  - Granada, Granada
  - A Coruña, La Coruña
  - Madrid, Madrid
  - Seville, Sevilla
  - Valencia, Valencia
- London, United Kingdom

REFERENCES:
- [Derived] Tong X, Le Pogam S, Li L, Haines K, Piso K, Baronas V, Yan JM, So SS, Klumpp K, Najera I. In vivo emergence of a novel mutant L159F/L320F in the NS5B polymerase confers low-level resistance to the HCV polymerase inhibitors mericitabine and sofosbuvir. J Infect Dis. 2014 Mar 1;209(5):668-75. doi: 10.1093/infdis/jit562. Epub 2013 Oct 23. PMID 24154738